CLINICAL TRIAL: NCT03066830
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin Added to a Sulfonylurea Alone or in Combination With Metformin in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on a Sulfonylurea Alone or With Metformin
Brief Title: Efficacy and Safety of Sotagliflozin Versus Placebo in Participants With Type 2 Diabetes Mellitus on Background of Sulfonylurea Alone or With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC14835; 2016-002826-35 (EudraCT Number); U1111-1186-2612 (Other: UTN)
Record Dates: First submitted 2017-02-24; First posted 2017-02-28 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin 400 mg (Experimental): Following a 2-week run-in phase, participants received two Sotagliflozin tablets of 200 mg, orally once daily, before the first meal of the day plus Metformin and Sulfonylurea as prescribed for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 79 weeks.
  Interventions: Drug: Sotagliflozin (SAR439954)
- Placebo (Placebo Comparator): Following a 2-week run-in period, participants were randomized to matching placebo administered as 2 tablets, once daily, before the first meal of the day plus Metformin and Sulfonylurea as prescribed for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 79 weeks.
  Interventions: Drug: Placebo; Drug: Metformin; Drug: Sulfonylurea

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Sotagliflozin 400 mg
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo
Drug: Sulfonylurea — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To demonstrate the superiority of Sotagliflozin 400 milligrams (mg) versus placebo on Hemoglobin A1c (HbA1c) reduction at Week 26 in participant with type 2 diabetes (T2D) who have inadequate glycemic control with a Sulfonylurea alone or in combination with Metformin.

Secondary Objectives:

* To compare Sotagliflozin 400 mg versus placebo based on:
* Change from baseline in fasting plasma glucose (FPG).
* Change from baseline in systolic blood pressure (SBP) for participants with baseline SBP ≥130 millimeter of mercury (mm Hg).
* Change from baseline in SBP for all participants.
* Change from baseline in body weight.
* Percentage of participants with HbA1c <6.5% and <7.0%.
* To evaluate the safety of Sotagliflozin 400 mg versus placebo throughout the 79-week trial.

DETAILED DESCRIPTION:
The duration per participants is up to 85 weeks, including a Screening Period consisting of a Screening phase of up to 2 weeks and a 2-week single-blind Run-in phase, a 26-week double blind Core Treatment Period, a 53 week double blind Extension, and a 2-week post treatment Follow-up period to collect safety information.

ELIGIBILITY:
Inclusion criteria :

* Participants with T2D treated with a Sulfonylurea (≥half the maximum recommended dose as per local label or maximum tolerated dose [documented]) as monotherapy or in combination with Metformin (≥1500 mg per day or maximum tolerated dose [documented]) each at a stable dose for at least 12 weeks without a dose adjustment before screening.
* Signed written informed consent.

Exclusion criteria:

* At the time of screening, age <18 years or < legal age of majority, whichever is greater.
* Body Mass Index (BMI) ≤20 or >45 kilograms per meter square (kg/m^2) at Screening.
* Hemoglobin A1c (HbA1c) <7% or HbA1c >10% via central lab test at screening.
* Fasting plasma glucose (FPG) >15 mmol/L (270 mg/dL) measured by the central laboratory at screening (Visit 1), and confirmed (>15 mmol/L [270 mg/dL]) by a repeat test before randomization.
* Women of childbearing potential with no effective contraceptive method.
* Treated with an antidiabetic pharmacological regimen other than a Sulfonylurea at a stable dose with or without Metformin within 12 weeks preceding the screening visit.
* Previous insulin use >1 month (at any time, aside from treatment of gestational diabetes).
* History of prior gastric surgical procedure including gastric banding or inflammatory bowel disease within 3 years before the Screening Visit.
* History of diabetic ketoacidosis or nonketotic hyperosmolar coma within 12 weeks prior to the Screening Visit.
* History of severe hypoglycemia within 6 months prior to the Screening visit.
* Systolic blood pressure (SBP) >180 millimeter per mercury (mmHg) or diastolic blood pressure (DBP) >100 mmHg or history of hypertensive emergency.
* Aspartate aminotransferase and/or alanine aminotransferase: >3 times the upper limit of the normal laboratory range (ULN).
* Total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome).
* Use of systemic glucocorticoids (excluding topical or ophthalmic, application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
* Pregnancy, breastfeeding.
* Participants is unwilling to perform self-monitoring of blood glucose (SMBG), and complete the participant's diary as required per protocol.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (76):
- United States (28):
  - Investigational Site Number 8403003, Litchfield Park, Arizona
  - Investigational Site Number 8403018, Peoria, Arizona
  - Investigational Site Number 8403009, Greenbrae, California
  - Investigational Site Number 8403012, Huntington Park, California
  - Investigational Site Number 8403019, Los Angeles, California
  - Investigational Site Number 8403034, Montclair, California
  - Investigational Site Number 8403016, Spring Valley, California
  - Investigational Site Number 8403014, Tustin, California
  - Investigational Site Number 8403001, Northglenn, Colorado
  - Investigational Site Number 8403029, Bradenton, Florida
  - Investigational Site Number 8403004, New Port Richey, Florida
  - Investigational Site Number 8403020, North Miami Beach, Florida
  - Investigational Site Number 8403026, Ocoee, Florida
  - Investigational Site Number 8403032, Orlando, Florida
  - Investigational Site Number 8403008, Palm Harbor, Florida
  - Investigational Site Number 8403006, Pembroke Pines, Florida
  - Investigational Site Number 8403013, Port Charlotte, Florida
  - Investigational Site Number 8403007, Nampa, Idaho
  - Investigational Site Number 8403011, Flint, Michigan
  - Investigational Site Number 8403025, Richfield, Minnesota
  - Investigational Site Number 8403021, Henderson, Nevada
  - Investigational Site Number 8403028, Greensboro, North Carolina
  - Investigational Site Number 8403015, Shelby, North Carolina
  - Investigational Site Number 8403033, Hatboro, Pennsylvania
  - Investigational Site Number 8403030, Kingsport, Tennessee
  - Investigational Site Number 8403002, Dallas, Texas
  - Investigational Site Number 8403022, Houston, Texas
  - Investigational Site Number 8403005, Burke, Virginia
- Bulgaria (3):
  - Investigational Site Number 1003003, Plovdiv
  - Investigational Site Number 1003002, Rousse
  - Investigational Site Number 1003004, Sofia
- Investigational Site Number 2333003, Pärnu, Estonia
- Hungary (11):
  - Investigational Site Number 3483001, Balatonfüred
  - Investigational Site Number 3483007, Budapest
  - Investigational Site Number 3483008, Budapest
  - Investigational Site Number 3483010, Budapest
  - Investigational Site Number 3483004, Budapest
  - Investigational Site Number 3483006, Budapest
  - Investigational Site Number 3483011, Gyula
  - Investigational Site Number 3483009, Hatvan
  - Investigational Site Number 3483005, Kecskemét
  - Investigational Site Number 3483003, Pécs
  - Investigational Site Number 3483012, Zalaegerszeg
- Poland (6):
  - Investigational Site Number 6163005, Gdansk
  - Investigational Site Number 6163006, Gdynia
  - Investigational Site Number 6163003, Katowice
  - Investigational Site Number 6163002, Poznan
  - Investigational Site Number 6163001, Warsaw
  - Investigational Site Number 6163004, Wroclaw
- Romania (2):
  - Investigational Site Number 6423004, Bucharest
  - Investigational Site Number 6423002, Iași
- Slovakia (6):
  - Investigational Site Number 7033006, Bratislava
  - Investigational Site Number 7033001, Bratislava
  - Investigational Site Number 7033002, Bratislava
  - Investigational Site Number 7033004, Malacky
  - Investigational Site Number 7033003, Štúrovo
  - Investigational Site Number 7033007, Trenčín
- South Korea (8):
  - Investigational Site Number 4103001, Goyang-Si, Gyeonggi-Do
  - Investigational Site Number 4103011, Guri-Si, Gyeonggi-Do
  - Investigational Site Number 4103003, Seongnam-Si, Gyeonggi-Do
  - Investigational Site Number 4103007, Seoul
  - Investigational Site Number 4103006, Seoul
  - Investigational Site Number 4103010, Seoul
  - Investigational Site Number 4103005, Seoul
  - Investigational Site Number 4103009, Wonju-Si, Gangwon-Do
- Ukraine (3):
  - Investigational Site Number 8043001, Kyiv
  - Investigational Site Number 8043003, Kyiv
  - Investigational Site Number 8043002, Kyiv
- United Kingdom (8):
  - Investigational Site Number 8263012, Birmingham
  - Investigational Site Number 8263009, Cardiff
  - Investigational Site Number 8263007, Glasgow
  - Investigational Site Number 8263008, Hexham
  - Investigational Site Number 8263003, Inverness
  - Investigational Site Number 8263014, Liverpool
  - Investigational Site Number 8263011, Manchester
  - Investigational Site Number 8263010, Reading

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) and supporting clinical documents are available for request at clinicalstudydatarequest.com. While making information available Sanofi continues to protect the privacy of the participants in clinical trials and to remove commercially confidential information (CCI). Details on Data Sharing criteria and process for requesting access can be found at this web address: clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 76 investigative sites in the United States, Bulgaria, Estonia, Hungary, Republic of Korea, Poland, Romania, Slovakia, Ukraine, United Kingdom from 24 February 2017 to 30 April 2019.
Pre-assignment Details: Participants with a diagnosis of Diabetes Mellitus were enrolled equally in 1 of 2 treatment groups, Sotagliflozin 400 milligrams (mg) and Placebo.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 400 mg
Started | 254 | 253
Completed | 221 | 231
Not Completed | 33 | 22
Not completed — At the Participant's own Request | 16 | 17
Not completed — Other | 3 | 0
Not completed — Poor Compliance to Protocol | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 11 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 254 | 253 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.9) | 63.3 (8.8) | 63.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 104 | 228
  Male | 130 | 149 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 53 | 96
  Not Hispanic or Latino | 210 | 198 | 408
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 28 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 8 | 16
  White | 211 | 215 | 426
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.18 (0.83) | 8.20 (0.83) | 8.19 (0.83)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 133.08 (14.21) | 134.30 (13.01) | 133.69 (13.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26
Description: Missing data are imputed using the retrieved dropouts imputation method. An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline to Week 26
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percentage HbA1c
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 254 | 253
percentage HbA1c | 0.06 (0.082) | -0.70 (0.068)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of Metformin use at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Square (LS) Mean = -0.76, 95% CI 2-sided [-0.946 to -0.574], Standard Error of Mean 0.095

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: Missing data are imputed using the retrieved dropouts imputation method. An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 254 | 253
millimole per liter (mmol/L) | 0.277 (0.2691) | -1.331 (0.1844)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of Metformin use at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline fasting plasma glucose as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.608, 95% CI 2-sided [-2.1685 to -1.0471], Standard Error of Mean 0.286

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) for Participants With Baseline SBP ≥130 mmHg
Description: Missing data are imputed using the washout imputation method under the missing, not at random framework. An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: Analysis was performed on ITT population in participants with baseline SBP ≥130 mmHg.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 146
mmHg | -3.58 (1.052) | -4.41 (1.061)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 12 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of Metformin use at screening and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.5172, ANCOVA; Difference in LS Means = -0.82, 95% CI 2-sided [-3.316 to 1.669], Standard Error of Mean 1.272

4. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants
Description: Missing data are imputed using washout imputation method under the missing not at random framework. An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: ITT population included all randomized participants .
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 254 | 253
mmHg | -0.69 (0.826) | -1.71 (0.830)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 12 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of Metformin use at screening, randomization strata of mean SBP (<130, ≥ 30 mmHg) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.2994, ANCOVA; Difference in LS Means = -1.02, 95% CI 2-sided [-2.946 to 0.907], Standard Error of Mean 0.983

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Missing data are imputed using the retrieved dropouts imputation method. An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 254 | 253
kilogram (kg) | -0.29 (0.206) | -1.70 (0.215)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of Metformin use at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.41, 95% CI 2-sided [-1.932 to -0.884], Standard Error of Mean 0.267

6. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 254 | 253
percentage of participants | 1.6 | 8.3
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Percentage difference between treatment groups using the Cochran-Mantel-Haenszel test stratified by the randomization strata of HbA1c (≤ 8.5, >8.5%) at screening, randomization strata of mean SBP (<130,≥130 mmHg) at screening, randomization strata of metformin use at the screening. Missing data at Week 26 were assigned a status of non-responder in the analysis; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Percentage difference = 6.7, 95% CI 2-sided [3.03 to 10.47]

7. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 254 | 253
percentage of participants | 8.7 | 26.1
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Percentage difference between treatment groups using the Cochran-Mantel-Haenszel test stratified by the randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization strata of Metformin use at screening. Missing data at Week 26 were assigned a status of non-responder in the analysis; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage difference = 17.4, 95% CI 2-sided [11.16 to 23.73]

8. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤ 70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤ 70 mg/dL]. Participants may be reported in more than one category.
Time Frame: Up to 79 weeks in the treatment period
Population: Safety population was defined as all randomized participants who had received at least 1 dose of the double-blind investigational medicinal product.
Measure: Number; unit: percentage of participants
Groups:
- Sotagliflozin 400 mg: Following a 2-week run-in phase, participants received two Sotagliflozin tablets of 200 milligrams (mg), orally once daily, before the first meal of the day plus Metformin and Sulfonylurea as prescribed for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 79 weeks.
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 253 | 254
percentage of participants
  Any hypoglycemia | 22.1 | 19.7
  Documented symptomatic hypoglycemia | 13.0 | 11.4
  Severe or documented symptomatic hypoglycemia | 13.0 | 11.8

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to 82.9 weeks) + 2 weeks
Description: Safety population included all randomized participants who received at least one dose of double-blind investigational medicinal product (IMP). One participant randomized to Placebo who was dosed with Sotagliflozin 400 mg treatment during the study and summarized in the Sotagliflozin 400 mg arm in the safety population.
Groups:
- Placebo: Following a 2-week run-in period, participants were randomized to matching placebo administered as 2 tablets, once daily, before the first meal of the day plus Metformin and Sulfonylurea as prescribed for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 79 weeks. One participant randomized to Placebo who was dosed with Sotagliflozin 400 mg treatment during the study is included in the Sotagliflozin 400 mg arm in the safety population.
- Sotagliflozin 400 mg: Following a 2-week run-in phase, participants received two Sotagliflozin tablets of 200 milligrams (mg), orally once daily, before the first meal of the day plus Metformin and Sulfonylurea as prescribed for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 79 weeks. One participant randomized to Placebo who was dosed with Sotagliflozin 400 mg treatment during the study is included in the Sotagliflozin 400 mg arm in the safety population.
Arm/Group | Placebo | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 2/253 | 2/254
Serious Adverse Events (participants affected / at risk) | 40/253 | 32/254
Other Adverse Events (participants affected / at risk) | 90/253 | 71/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=253) | Sotagliflozin 400 mg (N=254)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 2
Nerve compression (Nervous system disorders) | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0
Post stroke epilepsy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=253) | Sotagliflozin 400 mg (N=254)
Diarrhoea (Gastrointestinal disorders) | 11 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 48 | 14
Nasopharyngitis (Infections and infestations) | 23 | 21
Upper respiratory tract infection (Infections and infestations) | 19 | 9
Urinary tract infection (Infections and infestations) | 8 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03066830/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03066830/SAP_001.pdf